CLINICAL TRIAL: NCT04753853
Title: Effect of Infiltrative Treatment of Stromal Vascular Fraction in Patellar Tendinopathy
Brief Title: Stromal Vascular Fraction (SVF) Injection in the Treatment of Patellar Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lipo-Tend
Record Dates: First submitted 2021-02-12; First posted 2021-02-15 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Patellar Tendinitis; Tendinopathy; Patellar Tendinopathy
Keywords: stromal vascular fraction; patellar tendinopathy; injection
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Intervention Model Description: Interventional Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stromal Vascular Fraction injection (Experimental): intra- and peri-tendon ultrasound-guided injection of Stromal Vascular Fraction
  Interventions: Procedure: Stromal Vascular Fraction injection

INTERVENTIONS:
Procedure: Stromal Vascular Fraction injection — intra- and peri-tendon ultrasound-guided injection of Stromal Vascular Fraction

SUMMARY:
The aim of the study is the evaluation of clinical and radiological results after the treatment of patellar tendinopathy through the injection of autologous ultrasound-guided, intra- and peri-tendon stromal vascular fraction.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be treated according to the study protocol.

Every patients will undergo to a single peri- and intra- tendon injection with Autologous Stromal Vascula Fraction (SVF).

At baseline and at every follow-ups patients will be evaluated clinically and radiologically.

In particular, clinical evaluation and questionnaires will be performed at baseline, 1, 3, 6, 12 and 24 months visits, Ultrasound will be performed at baseline, 6 and 12 months visits. MRI will be performed at baseline and 6 months visits.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound or MRI signs of patellar tendon pathology

Exclusion Criteria:

* BMI > 30
* Patients suffering from: rheumatic diseases, diabetes, infectious processes, epilepsy, severe osteoporosis
* Patients undergoing intra-tendon infiltration of another substance within the previous 6 months;
* Patients who had patellar tendon surgery within the previous 12 months;
* Immunodepression
* On going systemic inflammatory diseases (stabilized outcomes of such diseases are not considered absolute contraindications).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Victorian Institute of Sport Assessment-Patella (VISA-P) questionnaire | 6 months
  VISA-P score is a questionnaire that assesses symptoms, simple tests of function, and the ability to play sports. It contains 8 questions about patellar tendinosis, max score for asymptomatic individual is 100; theoretical minimum is 0

SECONDARY OUTCOMES:
Victorian Institute of Sport Assessment-Patella (VISA-P) questionnaire | Baseline, 1, 3, 6, and 12 months (at 24 month the questionnaire will be performed by telephone)
  VISA-P score is a questionnaire that assesses symptoms, simple tests of function, and the ability to play sports. It contains 8 questions about patellar tendinosis, max score for asymptomatic individual is 100; theoretical minimum is 0
EuroQol Visual Analogue Scale (EQ-VAS) | Baseline, 1, 3, 6, and 12 months (at 24 month the questionnaire will be performed by telephone)
  EQ-VAS, which asks patients to indicate their overall health on a vertical visual analogue scale, ranging from "worst possible" to "best possible" health.
EQ-5D(EuroQol) | Baseline, 1, 3, 6, and 12 months (at 24 month the questionnaire will be performed by telephone)
  the EQ-5D profile, asks patients to classify their health based on self-assessed levels of problems ("no", "some", "extreme") on five dimensions.
Visual Analog Scale - VAS | Baseline, 1, 3, 6, and 12 months (at 24 month the questionnaire will be performed by telephone)
  Analogue scale represented by a line of 10 cm length, ranging from "absence of pain" to "the worst imaginable pain "
Tegner score | Baseline, 1, 3, 6, and 12 months (at 24 month the questionnaire will be performed by telephone)
  Tegner's activity scale classifies the activity according to work and sports activities on a scale from 0 to 10. Zero represents disability because of knee problems and 10 represents soccer a national or international level.
MRI evaluation | baseline and 6 month
  MRI performing and evaluation
ultrasound | baseline, 6 and 12 months
  ultrasound performing and thickness evaluation of the tendon

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy